CLINICAL TRIAL: NCT06309277
Title: A Two-Part Controlled Clinical Study to Evaluate Safety, Tolerability, Response, Pharmacokinetics and Pharmacodynamics of Single and Multiple Oral Doses of GM-1020 in Patients With Major Depressive Disorder
Brief Title: A Clinical Study to Evaluate of Single and Multiple Oral Doses of GM-1020 in Patients With MDD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilgamesh Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLG-100X
Record Dates: First submitted 2024-01-29; First posted 2024-03-13 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder
Keywords: MDD
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): GM-1020 (oral)
  Interventions: Drug: GM-1020
- Placebo (Placebo Comparator): Placebo (oral)
  Interventions: Drug: GM-1020

INTERVENTIONS:
Drug: GM-1020 — N-methyl-D-aspartate (NMDA) receptor antagonist

SUMMARY:
The aim of this Phase 2a study in patients with MDD is to assess safety and tolerability and preliminary antidepressant efficacy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patient is male or female, of any ethnic origin.
2. Patient is aged between 18 to 65 years, inclusive.
3. Patient has a body mass index (BMI) of 18.0 to 35.0 kg/m2, inclusive.
4. Patient is ≥50 kg.
5. Patient meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnostic criteria for recurrent MDD without psychotic features based on the Mini-International Neuropsychiatric Interview (MINI) at Screening. Comorbid anxiety disorders (e.g., social anxiety disorder, panic disorder, generalised anxiety disorder, specific phobia, agoraphobia) and cluster C personality disorders (avoidant, dependent and obsessive-compulsive) are allowed, provided that MDD is considered the primary diagnosis.
6. Current moderate to severe MDD as confirmed with a MADRS-SIGMA total score >22 and CGI-S score >3 at Screening and Day -1.
7. Patient is either not currently taking antidepressants (and hasn't for at least 6 weeks prior to Screening) or is being treated with an SSRI or SNRI antidepressant drug according to national guidelines during the current MDD episode.

   a. If the patient is currently being treated with SSRI or SNRI antidepressants, these have been prescribed at a stable dose and the dose has remained unchanged for at least 6 weeks prior to Screening. However, the following medications are not permitted during the study at any time: NMDA receptor antagonists (including ketamine, esketamine) and 5-HT2A receptor agonists (including psilocybin, DMT, 5-MeO-DMT). No augmentation strategies will be permitted.
8. Changes in current drug treatment or psychological treatment for depression are not foreseen for the duration of the study.

Key Exclusion Criteria:

1. Current or recent history of clinically significant suicidal ideation or behaviours as defined by:

   1. Suicidal ideation as endorsed on items 4 or 5 on the C-SSRS within 6 months prior to Screening, or
   2. Suicidal behaviours within 1 year prior to Screening, or
   3. Clinical assessment of significant suicidal risk. Patients with a prior suicide attempt of any sort, or prior serious suicidal ideation/plan >6 months ago, should be carefully screened for current suicidal ideation and only included at the discretion of the Investigator.
2. Involuntary psychiatric hospitalisation in the current episode. Previous involuntary psychiatric hospitalisation should be carefully considered and only included at the discretion of the Investigator.
3. Lifetime diagnosis of any DSM-5 psychotic disorders, bipolar or related disorders, post-traumatic stress disorder (PTSD), complex-PTSD and borderline personality disorder. Other psychiatric disorders besides MDD should not be the primary disorder.
4. Patient has failed previous treatment with rapidly acting antidepressant drugs, such as NMDA receptor antagonists (e.g., ketamine, esketamine) or 5-HT2A receptor agonists (e.g., psilocybin, DMT, 5-MeO-DMT) or neuromodulating treatments, such as electroconvulsive therapy, transcranial magnetic stimulation, vagus nerve stimulation, or deep brain stimulation.
5. Patient is currently or has recently (within 6 weeks prior to Day 1) been treated with antipsychotic medication.
6. Use of psychoactive substances (including ketamine, esketamine or psychedelics, excluding cannabis) during the 6 weeks prior to Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | Baseline, Day 42
  Clinical monitoring of safety data from AE reporting, 12-lead ECG, vital signs, clinical laboratory evaluations, emergence of suicidal thoughts and ideations (Columbia-Suicidal Severity Rating Scale) and sedation (Modified Observer's Assessment of Alertness and Sedation).

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) Change from baseline to 72 hours | Baseline, 72 hours
  MADRS total score, sum of 10 item scores (each on a 0 (best value) to 6 (worst value)scale), assesses the severity of depressive symptoms on a continuous scale from 0 (the best) to 60 (the worst).

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Marek, MD, Study Chair — Gilgamesh Pharmaceuticals
Locations (1):
- MAC Clinical Research, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No